CLINICAL TRIAL: NCT03020836
Title: Evaluating Effective Methods for Referral for Smoking Cessation Counseling and High Blood Pressure Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, David S. Friedman, Professor, Johns Hopkins University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NA_00089710
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Smoking Cessation
MeSH Terms: conditions — Hypertension; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertension patient referral (Other): Referral to primary care physician for hypertension control: Patients with uncontrolled hypertension were referred to a primary care physician for treatment.
  Interventions: Behavioral: Referral to primary care physician for hypertension control
- Smoking cessation patient referral (Other): Referral to smoking quit line: Patients that were current smokers were referred to the Maryland smoking cessation quit line if they were willing.
  Interventions: Behavioral: Referral to smoking quit line

INTERVENTIONS:
Behavioral: Referral to primary care physician for hypertension control — Referral to primary care physician for hypertension control
  Arms: Hypertension patient referral
Behavioral: Referral to smoking quit line — Referral to Maryland Tobacco/Smoking quit line for help with smoking cessation
  Arms: Smoking cessation patient referral

SUMMARY:
Investigators conducted a clinic-based study to determine the magnitude of uncontrolled hypertension and current smoking in eye doctor's offices and sought to determine if referral to care results in actions taken by the patient.

DETAILED DESCRIPTION:
Smoking and hypertension are two modifiable risk factors that are linked to highly prevalent chronic diseases such as diabetes and cardiovascular disease. The ophthalmology waiting room has the potential to be an effective point of intervention to provide referral to primary care in addition to health education on preventive health topics.

The investigators therefore, conducted a clinic-based study to determine the magnitude of uncontrolled hypertension and current smoking in eye doctor's offices and to determine if referral to care results in actions taken by the patient.

The investigators determined the proportion of patients who have elevated blood pressure. Patients were referred appropriately and the proportion of participants who followed the recommendation to meet with their primary care doctor for elevated blood pressure at 4-6 weeks and 8-10 weeks was determined. In addition, those who consented to be in the study and admitted to smoking cigarettes were offered smoking cessation assistance through a quit line. Investigators also followed up on cigarette smoking at 4-6 weeks and 8-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age presenting to the glaucoma service and general eye service at Wilmer Eye Institute.

Exclusion Criteria:

* Non-English speakers
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with elevated blood pressure | 1 day (at study clinic visit)

SECONDARY OUTCOMES:
Proportion of patients that are current smokers | 1 day (at study clinic visit)
Proportion of patients with elevated blood pressure that sought referral care | From study visit to 10 weeks after
Proportion of patients that were current smokers that sought referral quit line assistance | From study visit to 10 weeks after

IPD SHARING:
Plan to Share IPD: No